CLINICAL TRIAL: NCT04714879
Title: Modulation of Memory Consolidation in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Technische Universität Berlin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MemorySFB
Record Dates: First submitted 2018-12-14; First posted 2021-01-19 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Sleep
Keywords: memory consolidation

STUDY DESIGN:
Intervention Model Description: 7 experimental stimulation conditions (including sham stimulation) are tested in a randomized, counterbalanced, within-subject design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow oscillating transcranial direct current stimulation (so-tDCS) (Experimental): 7 experimental daytime naps with so-tDCS of different frequencies (fixed frequency of 0.75 Hz versus individually adapted frequency) and durations (5 min, 2 min, 30 sec) (Crossover assignment, applicable for each participant)
  Interventions: Other: Device: anodal tDCS
- Sham stimulation (Sham Comparator): sham so-tDCS during a daytime nap (Crossover assignment, applicable for each participant)
  Interventions: Other: Device: no stimulation

INTERVENTIONS:
Other: Device: anodal tDCS — anodal current modulated by an oscillatory component including a fixed (0,75 Hz) versus individually adapted so-tDCS frequency with three different stimulation durations (5 min, 2 min, 30 sec)
  Arms: Slow oscillating transcranial direct current stimulation (so-tDCS)
Other: Device: no stimulation — sham stimulation
  Arms: Sham stimulation

SUMMARY:
The goal of the present study is to optimize effects of slow oscillatory transcranial direct current stimulation (so-tDCS) on sleep physiology and memory consolidation in humans by combining computational and experimental human models in an iterative process. The investigator therefore works in cooperation with Prof. Dr. Klaus Obermayer (TU Berlin), who contributes computation models with the aim to mechanistically understand the impact of different perturbations on sleep-related electrophysiological features, and to subsequently optimize so-tDCS parameters for inducing SO and spindle activity.

DETAILED DESCRIPTION:
Sleep plays an active role in long-term consolidation of memories. Specifically, slow oscillations (SO, large amplitude waves <1 Hz) and sleep spindles (8-15 Hz), that can be measured by electroencephalography (EEG), appear to be critical for declarative memories. According to the "active system consolidation" account, newly encoded memories are reactivated during sleep, accompanied by sharp-wave ripple events (80-100 Hz) in the hippocampus, and redistributed to cortical long-term storage networks through a coordinated dialog between the hippocampus and neocortex. This dialog is supposedly mediated by a particular coupling between cortical SO and thalamo-cortical fast spindles (12-15 Hz), with spindles preferably occurring during SO up-phases, and hippocampal ripples grouped at the troughs of fast spindles. Slow spindles (8-12 Hz) are a separate kind of sleep spindle activity whose function in memory consolidation is less well understood.

Interventions targeting sleep parameters may not only make it possible to beneficially modulate a vital aspect of memory consolidation, i. e., sleep-dependent memory consolidation, but may also help to delineate which specific elements of the neural dynamics during sleep are crucial for successful consolidation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 50-80 years
* screened as healthy in a structured telephone interview

Exclusion Criteria:

* Mini Mental Status Examination scores below 24
* history of severe untreated medical, neurological, and psychiatric diseases
* sleep disorders
* alcohol or substance abuse
* brain pathologies identified on MRI scan
* intake of medication acting primarily on the central nervous system (e.g., antipsychotics, antidepressants, benzodiazepines, or any type of over-the-counter sleep-inducing drugs such as valerian),
* nonfluent German language abilities.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in EEG power (μV²) of the slow oscillation frequency band (0.5-1 Hz) following so-tDCS during sleep | up to 20 weeks
  Investigation whether 7 different protocols of anodal tDCS (including SHAM) lead to distinct changes in slow oscillation power
Changes in EEG power (μV²) of the sleep spindles frequency band (12-15 Hz) following so-tDCS during sleep | up to 20 weeks
  Investigation whether 7 different protocols of anodal tDCS (including SHAM) lead to distinct changes in sleep spindle power
Changes in cross-frequency coupling (resultant vector length) between slow oscillations and sleep spindles following so-tDCS during sleep | up to 20 weeks
  Investigation whether 7 different protocols of anodal tDCS (including SHAM) lead to distinct changes in coupling between slow oscillations and sleep spindles

SECONDARY OUTCOMES:
Sleep architecture | up to 20 weeks
  Proportion of time spent in different sleep stages (in %) during the entire nap and following so-tDCS
Changes in EEG power (μV²) of the delta frequency band (1-4 Hz) following so-tDCS during sleep | up to 20 weeks
  Investigation whether 7 different protocols of anodal tDCS (including SHAM) lead to distinct changes in delta power

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Floeel, Prof., Study Director — University Medicine Greifswald
Locations (1):
- University medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ladenbauer J, Khakimova L, Malinowski R, Obst D, Tonnies E, Antonenko D, Obermayer K, Hanna J, Floel A. Towards Optimization of Oscillatory Stimulation During Sleep. Neuromodulation. 2023 Dec;26(8):1592-1601. doi: 10.1016/j.neurom.2022.05.006. Epub 2022 Aug 16. PMID 35981956